CLINICAL TRIAL: NCT06732089
Title: Determining the Feasibility of Digital Interventions for Adults with Treatment-Resistant Depression
Brief Title: Digital Interventions for Adults with Treatment-Resistant Depression: a Pilot Study
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other); Toronto Metropolitan University (Other)
Responsible Party: Sponsor
Other Study IDs: 21-274; Miner's Lamp Foundation (Other: University of Toronto)
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder (MDD); Major Depressive Episode; Treatment-Resistant Major Depressive Disorder
Keywords: pilot study; digital health monitoring; wearable device; remote measurement-based care; treatment-resistant depression; observational study; feasibility study; electronic data capture
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- rTMS: Participants in this group are enrolled to recieve rTMS treatment as part of their clinical care in the Interventional Psychiatry Program.
- IVK: Participants in this group are enrolled to receive intravenous ketamine (IVK) treatment as part of their clinical care in the Interventional Psychiatry Program.
- ECT: Participants in this group are enrolled to receive electroconvulsive therapy (ECT) as part of their clinical care in the Interventional Psychiatry Program.

SUMMARY:
The goal of this observational study is to learn about remote mental health monitoring technology for adults with treatment-resistant depression. The main question it aims to answer is: are digital mental health monitoring tools (an electronic data capture platform and wearable device (e.g., smartwatch or smart-ring)) feasible to implement alongside clinical treatment for depression? The secondary aim of this study is to inform preliminary clinical parameters for larger, definitive studies.

Participants receiving neuropsychiatric treatment (repetitive transcranial magnetic stimulation, intravenous ketamine, or electroconvulsive therapy) as part of their regular medical care for treatment-resistant depression in the Interventional Psychiatry Program will have their clinical assessment data entered into a digital platform and will wear an accessory-based wearable device for the duration of treatment.

DETAILED DESCRIPTION:
This observational study with retrospective data analysis is conducted in patients with treatment-resistant depression (TRD) undergoing neuropsychiatric clinical treatment (rTMS, IVK, or ECT) in the Interventional Psychiatry Program (IPP) at St. Michael's Hospital. Participants will have scores from a self-report assessment of anxiety (GAD-7) and a self-report (PHQ-9) or clinician-administered (MADRS) assessment of depression completed as part of clinical care entered into the Research Electronic Database Capture (REDCap) web-based platform after each treatment session. This will facilitate retrospective analysis of mental health symptom change and treatment response over the course of treatment. Participants will also have the opportunity to wear an accessory-based wearable device (e.g., smartwatch or ring) throughout the course of treatment to passively capture physiological biometrics of physical and mental health (e.g., heart rate, temperature, sleep, activity). This two-year pilot study aims to recruit a total of 200 participants with TRD to retrospectively assess the feasibility and efficacy of integrating remote health sensing and monitoring platforms in psychiatric clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18+) who are capable of giving informed consent
* Patients meeting diagnostic criteria for major depressive disorder (MDD) without psychotic symptoms according to the DSM-5
* Currently experiencing a major depressive episode (MDE)
* Montgomery-Asperg Depression Rating Scale (MADRS) score greater than 20 at screening
* Patients meeting criteria for treatment-resistant depression (TRD): failure of 2 or more adequate trials of antidepressant therapy of adequate dose and duration during the current episode
* Enrollment in one of the treatment modalities (rTMS, IVK, or ECT) at the Interventional Psychiatry Program at St. Michael's Hospital, Unity Health Toronto
* Ownership of a smartphone (for participants using wearable devices)

Exclusion Criteria:

* Individuals without Internet access (required to access study platforms)
* Medication changes, aside from the treatment received through the IPP, one month (28 days) before screening, or during the entire duration of treatment (variable based on treatment arm)
* Participants who do not speak English fluently enough to successfully communicate study information, answer questions accurately, and/or obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults suffering from treatment-resistant depression (TRD) who are being treated in the Interventional Psychiatry Program at St. Michael's Hospital, Unity Health Toronto. Patients have a confirmed diagnosis of Major Depressive Disorder (MDD) and are experiencing a Major Depressive Episode (MDE) at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility | From Screening and Baseline Visit (Day 0) to last treatment day (approximately 2-8 weeks depending on treatment group)
  To determine the feasibility of using a web-based digital platform and wearable devices to collect active and passive data, respectively, among adults receiving clinical treatment for treatment-resistant depression. This will be measured by: number of recruitments (minimum threshold of 6-7 participants/month), recruitment rates (relative to invited patient-participants; minimum threshold of 80%), dropout rates (maximum threshold of 30%), reasons for dropout (qualitative), and data completion/adherence rates (minimum threshold of 70%).

SECONDARY OUTCOMES:
Longitudinal Changes in Symptom Presentation | From Screening and Baseline Visit (Day 0) to last treatment day (approximately 2-8 weeks depending on treatment group)
  To quantify changes in active (clinical symptoms) and passive (physiological) measures of physical (activity) and mental health (depression, anxiety, sleep) over time. Active data will focus on anxiety and depression symptoms across treatment, as reported on the GAD-7, PHQ-9, and MADRS. Passive data will focus on physiological biometrics (e.g., heart rate, respiration, step count, metabolic equivalency, body temperature, sleep staging, skin conductance response) captured by the wearable devices.
Predicting Treatment Response, Remission, and Relapse | From Screening and Baseline Visit (Day 0) to last treatment day (approximately 2-8 weeks depending on treatment group)
  To model and predict the likelihood of a patient achieving anxiety/depression treatment response (reduction greater than or equal to 50% on clinical assessment), remission (assessment score less than clinical threshold), and relapse (assessment score greater than clinical threshold after achieving remission) captured through active self-/clinician-administered assessments, based on longitudinal active and passive data.
Personalized Digital Phenotype Profiling (pDPP) | From Screening and Baseline Visit (Day 0) to last treatment day (approximately 2-8 weeks depending on treatment group)
  To construct pDPPs (a.k.a. digital fingerprints) for each participant based on longitudinal active and passive data. This will be achieved using machine learning (ML), artificial intelligence (AI), and advanced data analytic principles.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Srihar Krishnan, Ph.D., Peng., F.C.A.E., Study Chair — Toronto Metropolitan University; Dr. Wendy Lou, Ph.D., Study Chair — Dalla Lana School of Public Health, University of Toronto
Locations (1):
- St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parkington K, Aguilar RJ, Lee GH, Rueda A, Adamsahib F, Al-Hassan M, Famuditimi S, Menzies P, Lin Q, Lou W, Krishnan S, Bhat V. Digital health monitoring for adults with treatment-resistant depression: Observational feasibility study protocol. PLoS One. 2025 Oct 24;20(10):e0333484. doi: 10.1371/journal.pone.0333484. eCollection 2025. PMID 41134764